CLINICAL TRIAL: NCT04603612
Title: The Role of mRNA-based Urine Test (Xpert Bladder Cancer Monitor) in Predicting the Need for Second Look Biopsy After Transurethral Resection of Non Muscle-invasive Bladder Tumor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Amr Abdel-Lateif El-Sawy, Principal Investigator, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AE 181020
Record Dates: First submitted 2020-10-18; First posted 2020-10-27 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Bladder Cancer
Keywords: Repeat TURBT; Recurrence; mRNA
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NMIBC patients (Other): Patients with diagnosed bladder tumors seen the urology department (Urology and Nephrology Center, Mansoura University, Egypt) will be assessed for eligibility to the study and inclusion criteria. Patients who are meeting these criteria will be asked to participate in this prospective study and will be provided with an informed consent form. Study participants will be enrolled, and the appropriate scheduled procedures will be performed.
  Interventions: Procedure: Primary TURBT

INTERVENTIONS:
Procedure: Primary TURBT — As shown in (Fig. 1), all patients will be thoroughly evaluated by medical history and physical exam, laboratory investigations, abdominal pelvic ultrasound (US). Then, all patients will be managed by cystoscopy and initial complete TURBT. Patients with benign pathology, non-urothelial carcinoma or muscle invasive disease, will be excluded from the study.
  After 4-6 weeks, eligible patients will be appointed for repeat resection TURBT.

SUMMARY:
The Xpert BC Monitor is an mRNA-based urinary marker test for BC surveillance which measures the levels of five target mRNAs (ABL1, ANXA10, UPK1B, CRH and IGF2) from a voided urine sample by real-time RT-PCR. The Xpert BC Monitor automates and integrates sample processing, nucleic acid amplification, and the detection of target sequences.

The performance of Xpert BC monitor regarding its sensitivity and negative predictive value was shown to be considerably high reaching 84% and 93%, respectively. Moreover, this high sensitivity was maintained in low-grade (77%) and Ta tumors (82%). Xpert BC monitor is going to gain now a wide popularity among practitioners in surveillance of NMIBC patients due to its simplicity to do, reliability and reproducibility.

The investigators hypothesize that; Xpert BC monitor may be a useful tool in evaluation of patients, who are potentially candidates for repeat TURBT. It can refine the indications of repeat biopsy by exclusion of cases with negative test.

DETAILED DESCRIPTION:
Bladder cancer (BC) is a common cancer worldwide and one of the most expensive to manage. This disease accounts for 6-8% of all male malignancies and 2-3% in women. Non muscle invasive bladder cancer (NMIBC) represents about 70% to 80% of bladder cancer. Of these, 70 % present as T1, 20 % as Ta, and 10 % as carcinoma in situ (CIS).

Many NMIBCs are amenable to treatment with transurethral resection of bladder tumor (TURBT) alone. However, despite the therapeutic impact of TURBT, bladder cancer (BCa) recurrence rate can be as high as 75%.

The significant risk of residual tumor after initial TURBT of NMIBC lesion has been demonstrated in many studies. Persistent disease after resection of T1G3 tumors has been observed in nearly 33% to 53% of patients after TURB. Moreover, the tumor is often understaged by initial resection, so the likelihood that a T1 tumor has been understaged and muscle-invasive disease is detected by second resection ranges from 4% to 25%.

Treatment of a Ta, T1 high-grade tumor and a T2 tumor is completely different, so correct staging is therefore important. It has been demonstrated that a second TURBT in patients with T1G3 tumor can increase recurrence-free survival.

A second look TURBT is recommended in the following situations; 1- After incomplete initial TURBT. 2- If there was no muscle in the specimen after initial resection. 3- In all T1 tumors. 4- In all G3 tumors.

These findings lead to many studies which reported on the development of new methods to avoid residual tumor at initial resection as narrow band imaging versus white light imaging. However, such evolutions cannot omit the need for second resection.

Despite its valuable role in completion the diagnosis and proper risk categorization of NMIBC, Second look TURBT is still considered an accessory invasive procedure with more added surgical risks of anesthetic and surgical complication as bleeding and perforation. In addition, the cost issue of hospital stay and operating theatre is a major consideration. Recent studies are searching for a less invasive tool that can replace or at least refine the role of second look TURBT.

The Xpert BC Monitor is an mRNA-based urinary marker test for BC surveillance which measures the levels of five target mRNAs (ABL1, ANXA10, UPK1B, CRH and IGF2) from a voided urine sample by real-time RT-PCR. The Xpert BC Monitor automates and integrates sample processing, nucleic acid amplification, and the detection of target sequences.

The performance of Xpert BC monitor regarding its sensitivity and negative predictive value was shown to be considerably high reaching 84% and 93%, respectively. Moreover, this high sensitivity was maintained in low-grade (77%) and Ta tumors (82%). Xpert BC monitor is going to gain now a wide popularity among practitioners in surveillance of NMIBC patients due to its simplicity to do, reliability and reproducibility.

The investigators hypothesize that; Xpert BC monitor may be a useful tool in evaluation of patients, who are potentially candidates for repeat TURBT. It can refine the indications of repeat biopsy by exclusion of cases with negative test.

ELIGIBILITY:
Inclusion Criteria:

* 1. Ability to give informed consent. 2. Patients receiving complete resection of NMIBC during initial TURBT. 3. Patients with histopathologically NMIBC.

Exclusion Criteria:

* 1. Patients with history of previous radiotherapy or systemic chemotherapy. 2. Concomitant upper tract urothelial carcinoma (UTUC). 3. Post initial TURBT histopathology report showing any of the following;

  1. Benign histopathology
  2. Low risk NMIBC patients (single lesion, primary, Ta, G1)
  3. Muscle invasive UC
  4. Non urothelial carcinoma of the bladder
  5. CIS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Accuracy of Xpert monitor for detection of positive repeat TURBT | 2 years
  performance of Xpert BC monitor as a diagnostic tool for possible residual malignancy after initial TURBT by comparing the results obtained by pre-repeat TURBT Xpert BC urine test (Test of the study) with results of second look biopsy whether benign or malignant (Standard test).

CONTACTS AND LOCATIONS:
Overall Officials: Amr A Elsawy, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nephrology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Elsawy AA, Awadalla A, Abdullateef M, Ahmed AE, Abol-Enein H. Can repeat biopsy be skipped after initial complete resection of T1 bladder cancer? The role of a novel urinary mRNA biomarker. Urol Oncol. 2021 Jul;39(7):437.e11-437.e19. doi: 10.1016/j.urolonc.2021.02.009. Epub 2021 Mar 27. PMID 33785220